CLINICAL TRIAL: NCT02744209
Title: Immune Predictors of Response to Pembrolizumab Therapy in Stage IV Melanoma Patients
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Larry R. Pease, Professor of Biochemistry/Molecular Biology and Immunology, Mayo Clinic
Other Study IDs: 16-000531
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Stage IV Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma; RNA from leukocytes.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will test whether immune functions in individual cancer patients can be characterized in a quantitative manner using new technologies that analyze nucleic acids from peripheral blood cells and whether those quantitations can be used to predict the response outcomes of patients being treated with Pembrolizumab.

DETAILED DESCRIPTION:
The investigators will collect 50 milliliter blood samples from each patient before and after the first cycle of Pembrolizumab therapy. White blood cells will be separated according to cluster of differentiation (CD) markers into CD4+, CD8+, CD14+ populations using magnetic beads. A portion of each cellular fraction will be stimulated in the lab with a lineage-specific agonist cocktail. Ribonucleic acid (RNA) will be purified from both unstimulated and stimulated cell populations from both pre- and post-therapy timepoints for each patient. Lineage-specific transcriptomes will be quantitated and used to derive gene expression profiles for comparisons to clinical phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1 criteria to evaluate CT or PET(positron emission tomography)/CT assessments of tumor burden.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Hypersensitivity to pembrolizumab or any of its excipients.
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an agent against programmed cell death (PD)-1 (i.e., anti-PD-1) or a PD ligand (PD-L) (i.e.,anti-PD-L1 or anti-PD-L2).
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV melanoma
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Response to therapy | 12 weeks
  Patient response to therapy will be assessed using RECIST 1.1 criteria at 12 weeks. The investigators will use lymphocyte gene expression data to derive expression profiles that distinguish patients that respond to therapy (complete responses plus partial responses) from patients with disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Larry R Pease, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials